CLINICAL TRIAL: NCT04501341
Title: Effectivity and Safety of Autologous BM-MNC Stem Cell Therapy and Allogenic Umbilical Cord Mesenchymal Stem Cell for Type 2 Diabetes Mellitus Patients"
Brief Title: BM-MNC and UCMSC for Type 2 Diabetes Mellitus Patients
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Indonesia University (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. dr. Pradana Soewondo, SpPD-KEMD, Prof, Fakultas Kedokteran Universitas Indonesia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 132/PT02.FK25/U.Eu113/METEND/V
Record Dates: First submitted 2020-07-26; First posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-08

CONDITIONS: T2D
Keywords: type 2 diabetes; Bone-marrow mononuclear cells; Umbilical cord mesenchymal stem cells; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: 5 subjects receive BM-MNC and 10 subjects receive UC-MSC
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BM-MNC experimental (Experimental): Autologue bone marrow mononuclear cell
  Interventions: Biological: Bone-marrow aspiration, Intra-pancreatic Catheterisation of BM-MNC
- UC-MSC (Experimental): Umbilical cord mesenchymal stem cell
  Interventions: Biological: Intravenous Infusion of UC-MSC

INTERVENTIONS:
Biological: Bone-marrow aspiration, Intra-pancreatic Catheterisation of BM-MNC — Autologous bone-marrow mononuclear cells infused to the main blood vessels that supply the pancreas according to the results of previous pancreatic CT-scan, performed by interventional radiologist. The target is to distribute the BM-MNCs equally in all part of the pancreas. Dosage: 1 x 10^5 - 1 x 10^6 CD34 cells/kgBW
  Arms: BM-MNC experimental
Biological: Intravenous Infusion of UC-MSC — Allogeneic umbilical cord tissue-derived mesenchymal stem cells will be given via intravenous infusion. Dosage: 2 x 10^6 cells/kgBW, twice, with three months interval
  Arms: UC-MSC

SUMMARY:
The aim of this preliminary study is to evaluate the safety and efficacy of bone-marrow mononuclear cells (BM-MNCs) and umbilical-cord tissue-derived mesenchymal stem cells (UC-MSCs) administration in type 2 diabetes patients

DETAILED DESCRIPTION:
Type 2 diabetes (T2D) patients had peripheral insulin resistance accompanied by progressive pancreatic beta cell degeneration and dysfunction due to glucotoxicity and lipotoxicity. Several studies have shown that the immune system plays a significant role in the pathogenesis of T2D. Bone-marrow mononuclear cells (BM-MNCs) and umbilical-cord tissue-derived mesenchymal stem cells (UC-MSCs) via its immunomodulatory properties have the potential to improve insulin resistance condition and pancreatic beta-cells dysfunction thus improve the glycemic control and insulin requirement in T2D patients. In this pilot study, we plan to recruit 15 T2D patients with total daily dose of insulin >= 0.5 unit/kgBW/day to receive BM-MNCs (5 subjects) or UC-MSCs injections (10 subjects). These subjects will be closely followed up for 12 months for evaluation of primary and secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes patients on insulin therapy with or without oral hypoglycemic agents, with total daily dose of insulin >= 0,5 unit/kg body weight
* Stable HbA1C in the last six months (HbA1c <= 8.5%)

Exclusion Criteria:

* Type 1 diabetes mellitus
* eGFR < 45 mL/min/m2 (for BM-MNC)
* Liver disease (moderate- severe)
* Active infection
* Contrast hypersensitivity (for BM-MNC)
* History of Malignancy
* Acute coronary syndrome in last three months
* Coronary arterial diseases with significant stenosis and has not carried out revascularization
* Pregnancy (for women subjects)

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-03-14 (Actual); Primary Completion 2021-12-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Decreasing total daily dose of insulin (>= 30%) | Before intervention, 1st, 3rd, 6th, and 12th month after intervention
  After intervention, blood glucose level will be reported by the subjects on weekly basis. The insulin dose and/or oral medication will be adjusted accordingly.

SECONDARY OUTCOMES:
Increasing of C-peptide level | Before intervention, 1st, 3rd, 6th, and 12th month after intervention
  Measurements were obtained with mixed meal tolerance test
Decreasing of insulin resistance level | Before intervention, 1st, 3rd, 6th, and 12th month after intervention
  Measurement of HOMA-IR, calculated using fasting C-peptide and fasting plasma glucose formula
Immunology/inflammatory markers | Before intervention, 1st, 3rd, 6th, and 12th month after intervention
  Measurements of Interleukin-10 and TNF-alfa from serum and supernatant from PBMC stimulation
Adverse events | Up to 12 months after intervention
  Thrombosis, hemorrhage, and infection
HbA1c | Before intervention, 1st, 3rd, 6th, and 12th month after intervention
  Stable HbA1c or decreasing HbA1c (from baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

REFERENCES:
- [Background] Itariu BK, Stulnig TM. Autoimmune aspects of type 2 diabetes mellitus - a mini-review. Gerontology. 2014;60(3):189-96. doi: 10.1159/000356747. Epub 2014 Jan 22. PMID 24457898
- [Background] Tsai S, Clemente-Casares X, Revelo XS, Winer S, Winer DA. Are obesity-related insulin resistance and type 2 diabetes autoimmune diseases? Diabetes. 2015 Jun;64(6):1886-97. doi: 10.2337/db14-1488. PMID 25999531
- [Background] Campbell RK, Martin TM. The chronic burden of diabetes. Am J Manag Care. 2009 Sep;15(9 Suppl):S248-54. PMID 19817513
- [Background] Fery F, Paquot N. [Etiopathogenesis and pathophysiology of type 2 diabetes]. Rev Med Liege. 2005 May-Jun;60(5-6):361-8. French. PMID 16035295
- [Background] Wehbe T, Chahine NA, Sissi S, Abou-Joaude I, Chalhoub L. Bone marrow derived stem cell therapy for type 2 diabetes mellitus. Stem Cell Investig. 2016 Dec 6;3:87. doi: 10.21037/sci.2016.11.14. eCollection 2016. PMID 28066789
- [Background] Guan LX, Guan H, Li HB, Ren CA, Liu L, Chu JJ, Dai LJ. Therapeutic efficacy of umbilical cord-derived mesenchymal stem cells in patients with type 2 diabetes. Exp Ther Med. 2015 May;9(5):1623-1630. doi: 10.3892/etm.2015.2339. Epub 2015 Mar 9. PMID 26136869
- [Background] Estrada EJ, Valacchi F, Nicora E, Brieva S, Esteve C, Echevarria L, Froud T, Bernetti K, Cayetano SM, Velazquez O, Alejandro R, Ricordi C. Combined treatment of intrapancreatic autologous bone marrow stem cells and hyperbaric oxygen in type 2 diabetes mellitus. Cell Transplant. 2008;17(12):1295-304. doi: 10.3727/096368908787648119. PMID 19364067
- [Background] Bhansali A, Asokumar P, Walia R, Bhansali S, Gupta V, Jain A, Sachdeva N, Sharma RR, Marwaha N, Khandelwal N. Efficacy and safety of autologous bone marrow-derived stem cell transplantation in patients with type 2 diabetes mellitus: a randomized placebo-controlled study. Cell Transplant. 2014;23(9):1075-85. doi: 10.3727/096368913X665576. PMID 23561959
- [Background] Hu J, Li C, Wang L, Zhang X, Zhang M, Gao H, Yu X, Wang F, Zhao W, Yan S, Wang Y. Long term effects of the implantation of autologous bone marrow mononuclear cells for type 2 diabetes mellitus. Endocr J. 2012;59(11):1031-9. doi: 10.1507/endocrj.ej12-0092. Epub 2012 Jul 13. PMID 22814142
- [Background] Chao YH, Wu HP, Chan CK, Tsai C, Peng CT, Wu KH. Umbilical cord-derived mesenchymal stem cells for hematopoietic stem cell transplantation. J Biomed Biotechnol. 2012;2012:759503. doi: 10.1155/2012/759503. Epub 2012 Oct 3. PMID 23093863
- [Result] Weiss ARR, Dahlke MH. Immunomodulation by Mesenchymal Stem Cells (MSCs): Mechanisms of Action of Living, Apoptotic, and Dead MSCs. Front Immunol. 2019 Jun 4;10:1191. doi: 10.3389/fimmu.2019.01191. eCollection 2019. PMID 31214172
- [Result] Gao F, Chiu SM, Motan DA, Zhang Z, Chen L, Ji HL, Tse HF, Fu QL, Lian Q. Mesenchymal stem cells and immunomodulation: current status and future prospects. Cell Death Dis. 2016 Jan 21;7(1):e2062. doi: 10.1038/cddis.2015.327. PMID 26794657